CLINICAL TRIAL: NCT03805399
Title: Precision Treatment of Refractory Triple Negative Breast Cancer Based on Molecular Subtyping --FUSCC-TNBC- Umbrella Trial
Brief Title: FUSCC Refractory TNBC Umbrella (FUTURE)
Acronym: FUTURE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1807188-16
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Triple-negative Breast Cancer
Keywords: TNBC; Molecular Subtype; Precision Treatment; Umbrella
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pyrotinib; Capecitabine; 130-nm albumin-bound paclitaxel; camrelizumab; fluzoparib; apatinib; Sirolimus; Everolimus

STUDY DESIGN:
Intervention Model Description: The refractory mTNBC participants will be classified into four subtypes based on immunohistochemistry tests namely luminal androgen receptor (LAR), immunomodulatory (IM), basal-like immune suppressed (BLIS), and mesenchymal (MES).Then according to gene sequencing outcomes, different subtypes would receive different targeted therapy (combined with chemotherapy in three treatment arms).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- pyrotinib with capecitabine (Experimental): If patients were LAR subtype with HER2 gene activated mutation
  Interventions: Drug: Pyrotinib with Capecitabine
- AR inhibitor with CDK4/6 inhibitor (Experimental): If patients were LAR subtype without HER2 gene activated mutation, but had PIK3CA mutation, enter into arm B1; If patients were LAR subtype without HER2 gene activated mutation or PIK3CA mutation, enter into arm B2;If B2 was closed, enter into B4;
  Interventions: Drug: AR inhibitor combined with everolimus(B1) or CDK4/6 inhibitor(B2),or EZH2 inhibitor (B4)
- anti PD-1 with nab-paclitaxel (Experimental): If patients were IM subtype(CD8 positive T cell more than 20%)
  Interventions: Drug: anti PD-1 with nab-paclitaxel
- PARP inhibitor included therapy (Experimental): If patients were BLIS subtype and had a BRCA gene pathogenic mutation
  Interventions: Drug: PARP inhibitor included therapy
- BLIS with anti-VEGFR included therapy (Experimental): If patients were BLIS subtype and did not have a BRCA gene pathogenic mutation
  Interventions: Drug: BLIS with anti-VEGFR included therapy
- MES with anti-VEGFR included therapy (Experimental): If patients were MES subtype and without PI3K/AKT pathway activation
  Interventions: Drug: MES with anti-VEGFR included therapy
- mTOR inhibitor with nab-paclitaxel (Experimental): If patients were MES subtype and had PI3K/AKT pathway activation
  Interventions: Drug: mTOR inhibitor with nab-paclitaxel

INTERVENTIONS:
Drug: Pyrotinib with Capecitabine — If patients were LAR subtype with HER2 gene activated mutation, she would receive pyrotinib(EGFR-TKI) 400mg qd and capecitabine 1000mg/m2 bid (d1-d14)
  Other Names: SHR1258
  Arms: pyrotinib with capecitabine
Drug: AR inhibitor combined with everolimus(B1) or CDK4/6 inhibitor(B2),or EZH2 inhibitor (B4) — B1: if patients were LAR subtype without HER2 gene activated mutation, but had PI3KCA mutation, she would receive everolimus 10mg qd combined with AR inhibitor SHR3680 240mg qd continuously ; B2: if patients were LAR subtype without HER2 gene activated mutation or PI3KCA mutation, she would receive AR inhibitor SHR3680 240mg qd combined with CDK4/6 inhibitor SHR6390 150mg qd (three week on one week off); B4: If patients were LAR subtype without HER2 gene activated mutation or PI3KCA mutation, she would receive AR inhibitor SHR3680 240mg qd combined with EZH2 inhibitor SHR2554 300mg bid continuously
  Other Names: SHR3680 SHR6390
  Arms: AR inhibitor with CDK4/6 inhibitor
Drug: anti PD-1 with nab-paclitaxel — If patients were IM subtype, she will receive PD-1 antibody SHR1210 200mg q2w and nab-paclitaxel 100mg qw (three week on one week off).
  Other Names: SHR1210
  Arms: anti PD-1 with nab-paclitaxel
Drug: PARP inhibitor included therapy — If patients were BLIS subtype and had a BRCA gene pathogenic mutation, she will receive PARP inhibitor SHR3162 150mg bid and famitinib 20mg qd continuously .
  Other Names: SHR3162
  Arms: PARP inhibitor included therapy
Drug: BLIS with anti-VEGFR included therapy — If patients were BLIS subtype and did not have a BRCA gene pathogenic mutation , she will receive:
  E2: apatinib 250mg qd continuously combined with VP-16 50mg qd (three week on one week off); E3: famitinib 20mg qd continuously combined with VP-16 50mg qd (three week on one week off); E4: BP102 10mg/kg d1,d15 combined with nab-paclitaxel 100mg d1,d8,d,15; q4w
  Other Names: YN968D1
  Arms: BLIS with anti-VEGFR included therapy
Drug: MES with anti-VEGFR included therapy — If patients were MES subtype and without PI3K/AKT pathway activation,she will receive famitinib 20mg qd continuously combined with VP-16 50mg qd (three week on one week off).
  Other Names: YN968D1
  Arms: MES with anti-VEGFR included therapy
Drug: mTOR inhibitor with nab-paclitaxel — If patients were MES subtype and had PI3K/AKT pathway activation, she will receive mTOR inhibitor 10mg qd continuously combined with nab-paclitaxel 100mg qw (three week on one week off).
  Other Names: everolimus
  Arms: mTOR inhibitor with nab-paclitaxel

SUMMARY:
This is a Phase Ib/II, open-label, multi-center umbrella study evaluating the efficacy and safety of multiple targeted treatment in patients with refractory metastatic TNBC.The specific grouping of patients' depends on FUSCC 500+ gene panel testing and IHC subtype staining.

DETAILED DESCRIPTION:
This is a Phase Ib/II, open-label, multi-center,umbrella study evaluating the efficacy and safety of multiple targeted treatment in patients with metastatic TNBC who had disease progression during or following standard treatment with chemotherapy(anthracyclines,taxanes,platinums, vinorelbine,capecitabine,and gemcitabine included).300-400 patients will be screened and eligible participants will enter different treatment arms according to their molecular subtype (IHC staining) and FUSCC 500+ gene panel testing results. These tests would be done on their rebiopsy tumor specimen. Specifically, as to TNBC molecular subtyping,FUSCC data identified the genomic aberrations that drive each TNBC subtype by applying an integrative analysis combining somatic mutation, copy number aberrations (CNAs) and gene expression profiles, which classified TNBC patients into four subtypes, namely luminal androgen receptor (LAR), immunomodulatory (IM), basal-like immune suppressed (BLIS), and mesenchymal-like (MES). Then, FUSCC conducted a IHC subtyping model to replace complex genomic sequencing, which have been validated in FUSCC cohort.FUSCC 500+ gene panel was developed combining public database(TCGA, METABRIC, 560WES, MSKCC-IMPACT ect.) and FUSCC private TNBC database.New treatment arms may be added and/or existing treatment arms may be closed during the course of the study on the basis of ongoing clinical efficacy and safety as well as the current treatments available.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0, 1, or 2
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* Radiologic/objective evidence of recurrence or disease progression after available standard chemotherapy regimens(anthracyclines,taxanes, platinums, vinorelbine,capacitabine, and gemcitabine included) for metastatic breast cancer(MBC)
* Availability of a representative tumor specimen that is suitable for rebiopsy, IHC staining and gene sequencing
* Adequate hematologic and end-organ function, laboratory test results, obtained within 14 days prior to initiation of study treatment.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures as outlined for each specific treatment arm
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)
* have the cognitive ability to understand the protocol and be willing to participate and to be followed up.

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing CNS metastases
* Active or history of autoimmune disease or immune deficiency
* Significant cardiovascular disease
* History of malignancy other than breast cancer within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Treatment with chemotherapy, radiotherapy,immunotherapy or surgery (outpatient clinic surgery excluded)within3 weeks prior to initiation of study treatment.
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 3 years)
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)

SECONDARY OUTCOMES:
Disease Control Rate(DOR) | Baseline through end of study (approximately 3 years)
  Complete remission or partial remission or stable disease (according to RECIST1.1)
Progression Free Survival(PFS) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 3 years)
  time to progressive disease (according to RECIST1.1)
Overall Survival (OS) | Randomization to death from any cause, through the end of study (approximately 3 years)
  time to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin U Shao, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liu CC, Chen L, Cai YW, Chen YF, Liu YM, Zhou YJ, Shao ZM, Yu KD. Targeting EMSY-mediated methionine metabolism is a potential therapeutic strategy for triple-negative breast cancer. Cell Rep Med. 2024 Feb 20;5(2):101396. doi: 10.1016/j.xcrm.2024.101396. Epub 2024 Jan 29. PMID 38290515
- [Derived] Xiao Y, Ma D, Yang YS, Yang F, Ding JH, Gong Y, Jiang L, Ge LP, Wu SY, Yu Q, Zhang Q, Bertucci F, Sun Q, Hu X, Li DQ, Shao ZM, Jiang YZ. Comprehensive metabolomics expands precision medicine for triple-negative breast cancer. Cell Res. 2022 May;32(5):477-490. doi: 10.1038/s41422-022-00614-0. Epub 2022 Feb 1. PMID 35105939
- [Derived] Jiang YZ, Liu Y, Xiao Y, Hu X, Jiang L, Zuo WJ, Ma D, Ding J, Zhu X, Zou J, Verschraegen C, Stover DG, Kaklamani V, Wang ZH, Shao ZM. Molecular subtyping and genomic profiling expand precision medicine in refractory metastatic triple-negative breast cancer: the FUTURE trial. Cell Res. 2021 Feb;31(2):178-186. doi: 10.1038/s41422-020-0375-9. Epub 2020 Jul 27. PMID 32719455